CLINICAL TRIAL: NCT02579330
Title: Randomized Controlled Trial on Practicability of Coloshield in Transanal and Anal Surgery
Brief Title: Trial on Use of Coloshield in Transanal and Anal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daniel Steinemann, MD (Other)
Responsible Party: Sponsor-Investigator, Daniel Steinemann, MD, Sponsor-Investigator, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-341
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Fistula-in-ano; Rectal Polyp; Rectal Adenoma; Hemorrhoids; Anal Fissure
MeSH Terms: conditions — Rectal Fistula; Hemorrhoids; Fissure in Ano

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coloshield Group (Experimental): In the Intervention group the Coloshield Device (double balloon system) will be introduced at the beginning of surgery followed by a washout of the rectum with 500ml of saline solution. The grade of macroscopic contamination will be assessed.
  Interventions: Device: Coloshield; Other: Control
- Control Group (Sham Comparator): In the control Group the grade of macroscopic contamination will be assessed after rectal washout with 500ml of saline solution.
  Interventions: Other: Control

INTERVENTIONS:
Device: Coloshield — Coloshield is designed to occlude the rectum during surgery thus enabling the possibility for rectal washout and maintaining a clear operating field. The rod-shaped Instrument contains two silicon balloons which are inflated by means of a catheter. Several holes at the section in between the two balloons are connected to another catheter, which enable negative pressure to be established. By insufflation of the two balloons and establishment of a negative pressure between the balloons by means of connection to a closed drainage bottle the colon is occluded for the duration of surgery.
  Arms: Coloshield Group
Other: Control — In the control group no device is introduced but a rectal washout with 500ml of Saline solution in performed.

SUMMARY:
In various transanal and anal procedures it is desirable to clean the operating field from stool contamination. Thus mechanical bowel preparation is not well tolerated by patients. Enema does not provide sufficient effect. By the use of Coloshield a rectal washout might be performed and enable a clean operating field. In this randomized controlled trial the macroscopic contamination of the rectum with and without Coloshield is compared using the Boston Bowel Preparation Score (0-3).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for Fistula-in-ano, transanal resection of rectal Polyp or Adenoma, haemorrhoids or anal fissure.

Exclusion Criteria:

* Age <18 years
* inability to give informed consent
* pregnancy
* missing informed consent
* emergency Operation (<24hours of diagnosis and admission at emergency room)
* rectal strictures or Stenosis
* status post rectal resection or pelvic Radiation therapy
* inflammatory bowel disease with inclusion of the rectum
* need for mechanical bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Grade of macroscopic contamination according to adjusted Boston Bowel Preparation Score (0-3). | during initial surgery

SECONDARY OUTCOMES:
Stable position of Coloshield | during initial surgery
  The position of the deployed Coloshield at beginning of surgery and after 30 minutes is measured by rigid rectoscopy in cm from anal verge. Any slippage of the device during surgery is documented.
Injuries of the rectal mucosa | during initial surgery
  After removal of Coloshield by rigid rectoscopy any bleedings or tear injuries in the rectal mucosa (caused by Coloshield) are noted. It will be documented if there are bleedings or tear injuries or not, and if the exact number of bleedings and tear injuries.
Postoperative pain (VAS-score) | during hospitalisation (48h)
  The pain level on a VAS score from 0 (no pain) to 10 (strongest) 6 hours, 24 hours and 48 hours after surgery are documented.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Steinemann, MD, Principal Investigator — Cantonal Hospital Baselland, Switzerland
Locations (1):
- Kantonsspital Baselland, Department of Surgery, Bruderholz, Bruderholz, Switzerland

REFERENCES:
- [Derived] Cordewener C, Zurcher M, Muller PC, Muller-Stich BP, Zerz A, Linke GR, Steinemann DC. Randomized clinical trial on the use of a colon-occlusion device to assist rectal washout. Surg Endosc. 2021 Sep;35(9):5078-5087. doi: 10.1007/s00464-020-07992-9. Epub 2020 Sep 23. PMID 32968914